CLINICAL TRIAL: NCT04343014
Title: Effects of Tongue Root Retractor for Fibroscopic Intubation: a Feasibility Study
Brief Title: Tongue Root Retractor For Fibroscopic Intubation
Acronym: TRFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibroscopic intubation
Record Dates: First submitted 2017-10-08; First posted 2020-04-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Airway Management
Keywords: fibreoptic intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tongue Root Retractor (Experimental): Patients in this arm will receive fibroscopic endotracheal intubation with tongue root retractors.
  Interventions: Device: Tongue Root Retractor
- Conventional Fibroscope (Active Comparator): Patients in this arm will receive fibroscopic endotracheal intubation without any other devices.
  Interventions: Device: Conventional Fibroscope

INTERVENTIONS:
Device: Tongue Root Retractor — Fibroptic endutracheal intubation will be performed with tongue root retractor.
  Arms: Tongue Root Retractor
Device: Conventional Fibroscope — Fibroptic endutracheal intubation will be performed in conventional way.
  Arms: Conventional Fibroscope

SUMMARY:
Patients admit to the operation rooms of First Affiliated Hospital of Nanjing Medical University and requiring endotracheal intubation for general anesthesia will be enrolled in this case controlled study.

Patients 1) aged 18 to 70 years; 2) ASA graded I~II class; 3) general anesthesia should be performed under endotracheal intubation, will be included from this study. Patients 1) with organ transplant operations; 2) with thoracic and cardiac vascular surgery; 3) with severe heart or lung disease; 4) BMI over 35kg/m2, will be excluded from this study.

The primary aim is to compare airway clearance for fibreoptic tracheal intubation in each patient position. Secondary outcomes include times to view the vocal cord and carina, the time for tube advancement through the vocal cords, as well as the total time to achieve tracheal intubation.Two anesthesiologists with 5 years of experience in conventional endotracheal intubation and trained for fibreoptic intubation will perform the maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 70 years
* ASA graded I~II class
* scheduled for elective surgery requiring orotracheal intubation

Exclusion Criteria:

* with organ transplant operations
* with thoracic and cardiac vascular surgery
* with severe cadiac or pulmonary disease
* BMI over 35kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of intubation. | From start of intubation to successfully intubated (the endotracheal tube enters the trachea and the cuff is inflated), usually within 3 minutes.
  Successs of intubation at different attempts.

SECONDARY OUTCOMES:
Epiglottis level | within 30 seconds after the beginning of fibroscopy
  Airway clearance at the epiglottis level was assessed by observing whether the epiglottis was in contact with the posterior pharyngeal wall
Carina time | within 90 seconds
  time from the beginning of fibroscopy to the confirmation of the carina
Successful Intubation on 1st Attemp | from start of first intubation to end of first intubation attempt
  the success rate on 1st attempt
Number of attempts for tube advancement | within 120 seconds
  number of attempts for tube advancement from the beginning of fibroscopy to the success of the intubation

CONTACTS AND LOCATIONS:
Overall Officials: Zhengnian Ding, M.D., Study Chair — The First Affiliated Hospital with Nanjing Medical University; Xiaofei Cao, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Junbei Wu, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China